CLINICAL TRIAL: NCT01076218
Title: In Clinic Evaluation of the FreeStyle Navigator® Continuous Glucose Monitoring System Version 1.5
Brief Title: Navigator 1.5 Accuracy Study
Acronym: FSNQS
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC08-075
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2010-02

CONDITIONS: Diabetes Mellitus
Keywords: Continuous Glucose Monitoring; Accuracy; Continuous Glucose Error-Grid Analysis
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes: Patients with type 1 diabetes requiring multiple daily insulin injections or using insulin pumps
  Interventions: Device: FreeStyle Navigator Continuous Glucose Monitoring System Version 1.5

INTERVENTIONS:
Device: FreeStyle Navigator Continuous Glucose Monitoring System Version 1.5 — This is not an interventional study. Subjects must maintain their own diabetes treatment regimen throughout the study duration.

SUMMARY:
The purpose of the study is to confirm that the accuracy and safety of Version 1.5 of the FreeStyle Navigator Continuous Glucose Monitoring System are not impacted by the updates to the system algorithm and minor changes to the user interface and sensor delivery unit, such as adhesive sterilization method. It is anticipated that information collected will be submitted as a supplement to Premarket Approval Application (P050020) to the US Food and Drug Administration for approval to market this version of the system.

ELIGIBILITY:
Inclusion Criteria:

* History consistent with Type 1 diabetes for at least 2 years prior to enrollment;
* For at least 6 months prior to enrollment, insulin pump user or multiple daily insulin injections;
* At least 18 years of age;
* Available and capable of following the protocol instructions provided by the healthcare professional;
* Signed and dated Informed Consent form.

Exclusion Criteria:

* Pregnancy;
* Type 2, gestational, or secondary diabetes;
* Known allergy to medical grade adhesives or skin disinfectant;
* Skin abnormalities at the insertion sites that would confound the assessment of the effect of the device on the skin;
* Blood donation within 6 weeks prior to beginning study activities;
* Within past 6 months, severe hypoglycemic episode(s) resulting in hospitalization or loss of consciousness;
* Active myocardial ischemia;
* Previous history of stroke;
* Any other concomitant medical condition that in the opinion of the principal investigator would likely affect the evaluation of device performance and/or safety;
* Current participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 diabetes requiring multiple daily insulin injections or using an insulin pump
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara K Alva, Study Director — Abbott Diabetes Care
Locations (2):
- United States (2):
  - Diablo Clinical Research, Walnut Creek, California
  - Rainier Clinical Research, Renton, Washington